CLINICAL TRIAL: NCT07311460
Title: The Effects of High-intensity Interval Training on Selected Steroid Hormones and Psychological Features in Healthy Male Adolescents: A Randomized Controlled Trial
Brief Title: HIIT, Steroid Hormones and Mental Health in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: High Institute of Sports and Physical Education of Kef (Other)
Responsible Party: Principal Investigator, Nejmeddine Ouerghi, Principal Investigator, High Institute of Sports and Physical Education of Kef
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIIT-ADO-Stroid-H
Record Dates: First submitted 2025-11-20; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-11

CONDITIONS: Hormone
Keywords: adolescences; hormones; training period; mental health; physical performance
MeSH Terms: conditions — Psychological Well-Being | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training (HIIT) group (Experimental): The HIIT group performed a HIIT program consisting of three sessions per week for 10 weeks, including three sets of four to eight bouts of 30-second runs at high intensity (100-110% of maximal aerobic speed, MAS), interspersed with 30-second recovery runs at low intensity (50% MAS) between bouts.
  Interventions: Behavioral: High-intensity interval training (HIIT) program
- Control group (No Intervention): The participants in the control group maintained their normal daily activities.

INTERVENTIONS:
Behavioral: High-intensity interval training (HIIT) program — The HIIT program consisted of three sessions per week for 10 weeks, comprising of three sets of four to eight bouts of 30-s runs at high intensity [100-110% of maximal aerobic speed (MAS)], interspersed with 30-s recovery runs at low intensity (50% MAS) between bouts.
  Arms: High-intensity interval training (HIIT) group

SUMMARY:
The purpose of study was to investigate the effect of a high-intensity interval training (HIIT) intervention on cardiorespiratory fitness (CRF), hormonal, and mental health markers in male adolescents. The main question it aims to answer is: Does HIIT improve CRF, hormonal (testosterone and cortisol levels, testosterone:cortisol ratio), and mental health (depression, anxiety and stress scores) markers. Researchers will compare HIIT (designed to experimental group) to non-training intervention (designed to control group) to see if the training program works to improve the health status. HIIT consisted of three sessions per week for 10 weeks, comprising of three sets of four to eight bouts of 30-s runs at high intensity [100-110% of maximal aerobic speed (MAS)], interspersed with 30-s recovery runs at low intensity (50% of MAS) between bouts.

DETAILED DESCRIPTION:
High-intensity interval training (HIIT) is a time-efficient method for improving physical fitness in youth. However, limited evidence exists regarding its effects on testosterone and cortisol levels, testosterone:cortisol ratio, and mental health outcomes during adolescence, a critical period of development. This study was to investigate the effect of a HIIT intervention on cardiorespiratory fitness (CRF, expressed as maximal aerobic speed and maximal oxygen consumption), hormonal, and mental health markers in male adolescents. Twenty-eight healthy male adolescents (age, 14.9±0.74 yrs.) were randomized to a HIIT group (HIITG, n=15) or a non-training control group (CG, n=13). HIIT consisted of three sessions per week for 10 weeks, comprising of three sets of four to eight bouts of 30-s runs at high intensity [100-110% of maximal aerobic speed (MAS)], interspersed with 30-s recovery runs at low intensity (50% MAS) between bouts. Pre- and post-intervention assessments included CRF (VO2max), hormonal markers (testosterone, cortisol, and testosterone:cortisol ratio), and mental health markers (depression, anxiety and stress scores).

ELIGIBILITY:
Inclusion Criteria:

* male sex,
* age 14 to 16 years,
* normal weight according to the WHO child growth standards for BMI (BMI ≤ 85th percentile)
* parental approval.

Exclusion Criteria:

* medical conditions contraindicating intense physical exercise
* non-compliance with the training program
* habitual physical activity exceeding school physical education lessons
* current or recent (within 3 months) dietary supplementation or restriction
* incomplete data.

Ages: 14 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Male
Enrollment: 28 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
Testosterone | One day before the start and two days after the completion of the 10 weeks of training program.
  Testosterone concentration, expressed in nmol/L, was analyzed using enzyme-linked immunosorbent assay (ELISA) kits (Monobind, Inc., Lake Forest, CA).
Cortisol | One day before the start and two days after the completion of the 10 weeks of training program.
  Cortisol concentration, expressed in nmol/L, was analyzed using enzyme-linked immunosorbent assay (ELISA) kits (Monobind, Inc., Lake Forest, CA).
The testosterone/cortisol ratio | One day before the start and two days after the completion of the 10 weeks of training program.
  The testosterone/cortisol ratio (T/C) was calculated by dividing the testosterone value by the cortisol value for each participant.
Depression, Anxiety, and Stress Scale - 21 items (DASS-21) | Before the start and after the completion of the 10 weeks of training program.
  The DASS-21 is a self-report questionnaire that assesses symptoms of depression, anxiety, and stress (Lai et al., 2015). Each item is scored from 0 to 3, yielding a total score ranging from 0 to 63. Higher scores indicate worse psychological symptoms (greater levels of depression, anxiety, or stress). In the present study, we used the Arabic version of the DASS-21, which has been validated and shown to have good psychometric properties (Moussa et al., 2017), to ensure linguistic and cultural appropriateness for assessing adolescents' psychological well-being.

SECONDARY OUTCOMES:
Maximal aerobic speed | Before and after the 10 weeks of the training program.
  Maximal aerobic speed (MAS), expressed in km/h, was determined using the incremental running test (20-m shuttle run test) as previously described by (Léger et al. 1982). The test was designed to assess the aerobic capacity of schoolchildren, healthy adolescents, and adults.
Maximal oxygen consumption | Before and after the 10 weeks of the training program.
  Maximal oxygen consumption (VO2max), expressed in mL/kg/min, was determined using the incremental running test (20-m shuttle run test) as previously described by (Léger et al. 1982). The test was designed to assess the aerobic capacity of schoolchildren, healthy adolescents, and adults.

CONTACTS AND LOCATIONS:
Overall Officials: Nejmeddine Ouerghi, Ph.D, Principal Investigator — Research Unit "Sport Sciences, Health and Movement"(UR22JS01) High Institute of Sport and Physical Education of Kef, University of Jendouba, 7100 Kef, Tunisia.
Locations (1):
- Tunisia, El Kef, Boulifa, Tunisia

IPD SHARING:
Plan to Share IPD: No